CLINICAL TRIAL: NCT06599008
Title: Incidence and Pronostic of Junctional Rhythm After TAVI Implantation
Brief Title: Evaluate the Incidence of Junctional Rhythms Occurring During Post-procedure TAVI Hospitalization.
Acronym: JUNCTAVI
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: RNI 2024 MASSOULLIE; 2024-A01132-45 (Other: ANSM : Agence Nationale de Sécurité du Médicament et des Produits de Santé); 24.03051.000665 (Other: CPP: Comité de Protection des Personnes Ile de France III)
Record Dates: First submitted 2024-09-12; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Incidence of Junctional Rhythm
Keywords: Transcatheter Aortic Valve Implantation; Junctional rhythm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Transcatheter Aortic Valve Implantation (TAVI) aims to treat patients with symptomatic narrowing of the aorta by implanting an aortic bioprosthesis. This technique, which is currently highly developed, can lead to the appearance of cardiac conduction disorders following implantation, and in particular the presence of a junctional rhythm. Junctional rhythms are tachycardias involving a circuit between the atria and the ventricles (junction between the two compartments atrium and ventricle).

The goal of this observational study is to describe the incidence and pronostic of this rhythm disorder (junctional rhythm) following the TAVI procedure.

DETAILED DESCRIPTION:
Monocentric observational study including all patients implanted with aortic bioprosthesis [undergoing Transcatheter Aortic Valve Implantation (TAVI)] at Clermont-Ferrand University Hospital, between December 1st, 2023 and March 1st, 2025. Telemetric monitoring and daily electrocardiograms were used to identify junctional rhythms. The primary endpoint was pacemaker (PM) implantation between day 0 and day 30 after TAVI. Patients with a junctional rhythm at the time of hospitalization were recalled to find out whether they had benefited from PM implantation within 30 days after the TAVI procedure.

ELIGIBILITY:
Inclusion Criteria:

* Major patients who have undergone or are undergoing a TAVI procedure (since 01/12/2023) and who present a junctional rhythm.

Exclusion Criteria:

* Minor patients
* Patients already implanted with a pacemaker
* Atrial fibrillation
* Pregnant women.
* Patients under guardianship or legal protection
* Patients deprived of liberty
* Patients refusing to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients implanted with aortic bioprosthesis [undergoing Transcatheter Aortic Valve Implantation (TAVI)] at Clermont-Ferrand University Hospital, between December 1st, 2023 and March 1st, 2025. Telemetric monitoring and daily electrocardiograms were used to identify junctional rhythms.
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2024-10-05 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
The occurrence of junctional rhythm during hospitalization after TAVI procedure. | 30 days post TAVI procedure
  The primary endpoint was pacemaker (PM) implantation between day 0 and day 30 after TAVI. Patients with a junctional rhythm at the time of hospitalization were recalled to find out whether they had benefited from PM implantation within 30 days after the TAVI procedure.

SECONDARY OUTCOMES:
Describe the prognosis of the occurrence of a junctional rhythm during hospitalization following a TAVI procedure. | 30 days post TAVI procedure
  Need for pacemaker implantation between D0 and D30, following the TAVI procedure.
Investigate the association between the presence of a junctional rhythm following TAVI procedure and all-cause or cardiovascular mortality, rehospitalization, and heart failure. | 30 days post TAVI procedure
  Assessment of the prognosis of junctional rhythms: collection of all-cause mortality, cardiovascular mortality, presence of syncope, conduction disorder on Holter ECG, rehospitalizations, occurrence of heart failure at day 30 post TAVI.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Centre Hospitalier Universitaire de Clermont-Ferrand, Clermont-Ferrand
  - CHU clermont-Ferrand, Clermont-Ferrand

IPD SHARING:
Plan to Share IPD: No